CLINICAL TRIAL: NCT03425916
Title: Changes in Abdominal Muscles Performance and Inter-rectus Distance in Postpartum Women: an Ultrasonography and Electromyographic Study.
Brief Title: Changes in Abdominal Muscles Performance in Postpartum Women.
Status: Completed | Type: Observational
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Beatriz Arranz Martin, Physiotherapist, University of Alcala
Other Study IDs: BAM2018
Record Dates: First submitted 2018-01-25; First posted 2018-02-08 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Recti Diastasis; Pregnancy Related
Keywords: Hypopressive exercises; Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primiparous women: Women after normal, not operative, vaginal one-child delivery
  Interventions: Other: Physical therapy intervention
- Nulliparous women: Women without any child or pregnancy, age-matched

INTERVENTIONS:
Other: Physical therapy intervention — Primiparous women start a physical therapy intervention in week 6 after normal one-child delivery, based on abdominal and pelvic floor exercises, education and behavior advices. Abdominal muscle condition and activation are measured by transabdominal ultrasound and surface electromiography. This group is going to be examined after treatment and 6 and 12 months after treatment.
  Groups: Primiparous women

SUMMARY:
To describe and compare abdominal muscles and inter-rectus distance conditions in postpartum period in comparison with nulliparous women. Also to describe the activation changes during different abdominal exercises.

DETAILED DESCRIPTION:
Pregnancy and childbirth cause corporal changes in women, altering the structure and function of the abdominal and pelvic floor muscles. The distension of the muscular tissue and the possible diastasis recti can alter the performance of the abdominal musculature in the control of intra-abdominal pressure and the lumbo-pelvic stabilization in postpartum term. Abdominal exercise is highly recommended to restore these changes but there is not enough evidence about the effects of exercise modalities.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women
* Normal not operative delivery
* One child delivery

Exclusion Criteria:

* Two or more previous gestation
* Previous abdominal surgery
* Systemic disease, neurologic or metabolic disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primiparous women after normal, not operative, vaginal one-child delivery, recruited 6-7 weeks after delivery from Hospital Universitario Principe de Asturias (Alcala de Henares, Madrid)
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2019-05-06 (Actual)

PRIMARY OUTCOMES:
Inter-rectus distance (mm) | 1 day
  Inter-rectus abdominis distance in mm in rest position.

SECONDARY OUTCOMES:
Cross-sectional area (mm) | 1 day
  Cross-sectional area of rectus abdominis, external oblique, internal oblique and transversus abdominis in rest position.
Neuromuscular activity (mV) | 1 day
  Neuromuscular activity (mV) of rectus abdominis, external oblique and internal oblique + transversus abdominis in rest position.
Inter-rectus distance (mm) during an hypopressive exercise | 1 day
  Inter-rectus distance (mm) during an hypopressive exercise performance in supine position.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Torres, PhD, Study Director — University of Alcala
Locations (1):
- Beatriz Arranz Martin, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No